CLINICAL TRIAL: NCT03977246
Title: The Effect of an Open-placebo Intervention on Cycling Time-trial Performance
Brief Title: Effect of Open-placebo Intervention on Cycling Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OpenPlaceboCycling
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Exercise Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open-placebo (Experimental): The open-placebo intervention session
  Interventions: Behavioral: Open-placebo
- Control (Placebo Comparator): The control session
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Open-placebo — Application of the open-placebo intervention
  Arms: Open-placebo
Behavioral: Control — Application of the control session
  Arms: Control

SUMMARY:
This study evaluates the effect of an open-label placebo intervention on cycling time-trial performance.

DETAILED DESCRIPTION:
This study investigated the effect of open-placebo on cycling time-trial (TT) performance. Twenty-eight trained female cyclists completed a 1-km cycling TT following a control session or an open-placebo intervention. The intervention consisted of an individual presentation, provided by a medic, in which the concept of open-placebo was explained to the participant, before she ingested two red and white capsules containing flour; 15 min later, they performed the TT. In the control session, the participant sat quietly for 20 min.

ELIGIBILITY:
Inclusion Criteria:

* Females aged between 18 and 45 years old;
* A minimum of one-year training experience in cycling.

Exclusion Criteria:

* Smokers
* Chronic disease
* Prior or current use of steroids
* Use of creatine in the last 6 months
* Use of beta-alanine in the last 6 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Exercise performance | 20-min following open-placebo intervention
  Change in 1 km cycling time-trial performance

SECONDARY OUTCOMES:
Blood lactate | Immediately post-exercise
  Change in blood lactate concentration

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gualano, PhD, Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - University of Sao Paulo, São Paulo
  - School of Physical Education and Sport - USP, São Paulo

IPD SHARING:
Plan to Share IPD: No